CLINICAL TRIAL: NCT06926725
Title: Combined Effect of High Intensity Interval Training and Ultrasound Cavitation on Lipid Profile in Type 2 Diabetes Patients With Abdominal Obesity
Brief Title: Effect of High Intensity Interval Training and Ultrasound Cavitation on Lipid Profile in Type 2 Diabetes Patients
Acronym: Diabeties
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahmoud Awad Ramadan Elkholy (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Awad Ramadan Elkholy, lecturer of physical therapy, Beni-Suef University
Organization: Beni-Suef University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FPTBSUREC/0803/1241124
Record Dates: First submitted 2025-04-06; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet

STUDY DESIGN:
Intervention Model Description: Type two diabetic patients with abdominal obesity , randomly assigned into 3 equal groups: 66 patients
  1. study group (A) 22 patients : They will receive ultrasound cavitation , HIIT and diatery advice .
  2. study group (B) 22 patients : They will receive HIIT and diatery advice .
  3. control group 22 patients They will only receive diatery advice.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- group A (Experimental): 22 patients : They will receive ultrasound cavitation , HIIT and diatery advice .
  Interventions: Device: Cavitation : Study group A only will receive one session per week for three months (total 12 sessions ). Ultrasound treatments are performed using an applicator head with diameter 7 cm . Intensity :; Other: high intenisty exercise; Dietary Supplement: Diet
- Group B (Experimental): 22 patients : They will receive HIIT and diatery advice .
  Interventions: Other: high intenisty exercise; Dietary Supplement: Diet
- Group C (Placebo Comparator): 22 patients They will only receive diatery advice.
  Interventions: Dietary Supplement: Diet

INTERVENTIONS:
Device: Cavitation : Study group A only will receive one session per week for three months (total 12 sessions ). Ultrasound treatments are performed using an applicator head with diameter 7 cm . Intensity : — Cavitation :
  Study group A only will receive one session per week for three months (total 12 sessions ).
  Ultrasound treatments are performed using an applicator head with diameter 7 cm .
  Intensity : 0.1-0.5 w/cm2 (low) Frequency : 30-40 KHZ (low) Duration : 30 minutes
  Arms: group A
Other: high intenisty exercise — type: alternate high intensity exercise (aerobic or strength training) with recovery stages Intensity: high intensity (75%-95% HRmax) or RPE(14-16 hard to very hard ) ( according to patient tolerance), followed by active or passive recovery stage (30%-60% HRmax) or RPE(7-11 extremely light to light) .
  frequency : 3 days per week for three months (with no more than 2 consecutive days between sessions) Duration: 10 seconds to 4 minutes high intensity ,12 seconds to 5 minutes active or passive recovery .(according to patient tolerance) 5 minutes warm up pre exercise . 5 minutes cool down post exercise . Progress gradually. total duration :20-40 minutes (according to patient tolerance and progression)
  Arms: Group B; group A
Dietary Supplement: Diet — In all groups (both study groups A&B and control group).

SUMMARY:
The study aim to find out the combined effect of high intensity interval training and ultrasound cavitation on lipid profile in type two diabetic patient with abdominal obesity.

DETAILED DESCRIPTION:
study aim to find out the combined effect of high intensity interval training and ultrasound cavitation on lipid profile in type two diabetic patient with abdominal obesity.Type two diabetic patients with abdominal obesity , randomly assigned into 3 equal groups: 66 patients

1. study group (A) 22 patients : They will receive ultrasound cavitation , HIIT and diatery advice .
2. study group (B) 22 patients : They will receive HIIT and diatery advice .
3. control group 22 patients They will only receive diatery advice.

ELIGIBILITY:
Inclusion Criteria:

* patient with type 2 diabetes.
* waist circumference >102 cm in male ,>88 cm in female
* lipid profile range will be (between border line and high risk ).

Exclusion criteria:

Kidney disease Heart disease Lung disease ,Liver disease ,Neurological disorders ,Pregnant women , breast feeding, immune deficiency , cancer Heavy smoker

Exclusion Criteria:

-

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-04-11 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Anthropometric Measurements | 3 months
  It will be performed before and after the treatment . Weight in (kg) is measured by in body scale During the measurement of height in( cm) patient is barefoot . Body mass index (BMI): weight (kg)/ [ height (m)] 2
Lipid profile | 3 months
  contains (cholesterol, triglycerides, Low-density lipoprotein cholesterol (LDL), and high-density lipoprotein cholesterol (HDL)).

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-Suif University Hospital, GIZA, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
patient privacy ,confidentially and security concern

REFERENCES:
- [Background] Birendra Kumar Jha, Raman Mishra, Jitendra Kumar Singh, Satyam Prakash, & Kamlesh Kumar Yadav. (2024). Assessment of glycemic control and correlation of HbA1c level with lipid profile and duration of diabetes in type 2 diabetes mellitus patients. Janaki Medical College Journal of Medical Science, 12(02), 13-24. https://doi.org/10.3126/jmcjms.v12i02.68365
- See also: Related Info — https://doi.org/10.3126/jmcjms.v12i02.68365